CLINICAL TRIAL: NCT02266446
Title: Phase 1 Open Trial of Attention and Interpretation Modification (AIM) for Anxiety Disorders in Primary Care
Brief Title: Developing a Low-Intensity Primary Care Intervention for Anxiety Disorders
Acronym: AIM-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Memorial Hospital of Rhode Island (Other); Mclean Hospital (Other)
Responsible Party: Principal Investigator, Risa B Weisberg, Principal Investigator, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1308000908; 1R34MH097820-01A1 (NIH)
Record Dates: First submitted 2014-07-15; First posted 2014-10-17 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Anxiety Disorders
Keywords: anxiety disorders; cognitive bias modification; primary care; attention; interpretation; computer
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Attention & Interpretation Modification (Experimental): The final product will be web-delivered, so it may be completed at the clinic or home. Treatment will consist of 8, 30-minute, twice-weekly sessions designed to: a) decrease attention bias to threat and b) extinguish threat interpretations/reinforce benign interpretations of ambiguity. Attention bias will be modified via a dot probe task that increases attentional control by directing attention away from threat faces via probe location. Patients will complete 256 trials per session. Interpretation bias will be modified via a word-sentence association task which provides positive feedback when participants endorse benign interpretations of ambiguous sentences and negative feedback for threat interpretations. Participants will complete 150 training trials per session
  Interventions: Behavioral: Attention & Interpretation Modification

INTERVENTIONS:
Behavioral: Attention & Interpretation Modification
  Other Names: AIM; Cognitive Bias Modification

SUMMARY:
The purpose of the study is to develop a personalized, user-friendly computerized treatment for anxiety disorders linked to primary care. The computerized treatment is a type of Cognitive Bias Modification, which targets attention and interpretation biases known to maintain anxiety disorders.

DETAILED DESCRIPTION:
The primary goals of our 3-year, 2-phase project are to develop AIM for primary care linkage and assess its feasibility and acceptability. This protocol description only pertains to Part A (treatment development) and B (open trial).

As it is essential that AIM is eventually implementable in practice settings, we integrate implementation methods in our early development work. We will develop AIM to meet an existing need (low-intensity anxiety disorder treatment), ensure that it fits our local setting, and identify eventual implementation barriers and facilitators via an open pilot trial. We will strive to develop and pilot AIM in a manner that is perceived as compatible with existing practices, simple to use, advantageous relative to existing practice, and beneficial. In order to conduct ongoing evaluation, a team of "end users," including Primary Care Physicians (PCPs), nurses, patients and practice leaders at the Family Care Center (FCC) of Memorial Hospital of Rhode Island, our study site, and at other sites in Rhode Island and Massachusetts, will participate on an Advisory Panel (AP).

Part A: develop AIM including a: 1) personalization computer program that will create an idiographic stimulus set for each participant to be used in the treatment; 2) self-administered, personalized, Cognitive Bias Modification treatment; and 3) protocol for primary care linked delivery.

Part B: an open trial of AIM comprising 3 iterations of 6 patients each. After each iteration, our study team and the AP will review data on feasibility and acceptability of AIM and delivery methods, and make revisions as needed. 8 primary care patients with primary Generalized Anxiety Disorder, Social Anxiety Disorder, and/or Panic Disorder (with or without Agoraphobia) will be enrolled, in 3 iterations. Full assessments will occur pre- and post-treatment. Weekly measures of anxiety and depression will be collected, as will feedback from patients and PCPs about the research and delivery procedures. At the end of the 1st iteration (n=6), the research team and AP will discuss and compare our actual data to the target outcomes. Target outcomes were chosen on face validity, clinical experience, and, when available, relevant literature (e.g., efficacy target based on previous trials and what we deemed clinically meaningful change for low-intensity treatment). Deviations from target outcomes will prompt investigation and discussion, and possible revision of AIM or of research procedures. After revision, we will recruit 6 new patients for the 2nd iteration. At the end of this iteration, the team and AP will review data and make changes as needed. We will repeat this process in the 3rd iteration (n=6).

Part C will include a randomized controlled trial of the final protocol.

ELIGIBILITY:
Inclusion Criteria:

* Study site patient
* Age ≥18
* Primary diagnosis of Generalized anxiety disorder (GAD), Social Phobia (SP), and/or panic disorder with or without agoraphobia (PD/A)
* At least moderate anxiety severity (GAD-7 score > 10)
* English-speaking
* If on psychopharmacotherapy, stable dose for 3 months; to minimize learning effects, patients taking benzodiazepines will complete AIM prior to their first dose of the day
* No current psychotherapy
* No current severe psychiatric symptoms requiring immediate attention (e.g., imminent suicidality, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | 6-8 weeks after first treatment session

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7-Item Scale | 6-8 weeks after first treatment session
Patient Health Questionnaire-9 | 6-8 weeks after first treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Risa B Weisberg, PhD, Principal Investigator — Alpert Medical School of Brown University; Courtney Beard, PhD, Principal Investigator — Harvard Medical School/McLean Hospital
Locations (1):
- Family Care Center of Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States